CLINICAL TRIAL: NCT00885196
Title: A Double Blind, Randomized, Placebo Controlled, Multicenter, Dose Finding Study of Oral AEB071 Assessing Psoriasis Area and Severity Index (PASI) Response and a Function of Dose and Treatment Duration (Primary Outcome) in Patients With Plaque Psoriasis
Brief Title: A Dose Finding Study of AEB071 Assessing Psoriasis Area and Severity Index in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAEB071C2201; EUDRACT number: 2007-007160-19
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2016-04

CONDITIONS: Moderate and Severe Plaque Psoriasis
Keywords: Psoriasis; plaque psoriasis; inflammatory skin disease; scaly patches; AEB071
MeSH Terms: conditions — Lymphoma, Follicular; Psoriasis; Dermatitis | interventions — sotrastaurin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- AEB071 200 mg BID (Experimental)
  Interventions: Drug: AEB071
- AEB071 400 mg OD (Experimental)
  Interventions: Drug: AEB071
- AEB071 300 mg BID (Experimental)
  Interventions: Drug: AEB071
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo BID
Drug: AEB071
  Arms: AEB071 200 mg BID; AEB071 300 mg BID; AEB071 400 mg OD

SUMMARY:
This study is designed to provide efficacy and safety data of several doses of AEB071 so that the optimal dose and treatment duration can be chosen for testing in later studies in patients with plaque psoriasis (with a disease severity such that systemic treatment is justified). The treatment free Follow-up Period is designed to provide additional safety data and information on disease recurrence after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and Severe Plaque psoriasis diagnosed for at least 12 months (with or without psoriatic arthritis as comorbidity)that requires systemic therapy
* Severity of disease meeting all of the following three criteria:

  * PASI score of 10 or greater
  * Total Body Surface Area (BSA) affected by plaque psoriasis of 10% or greater
  * Investigator's Global Assessment (IGA) score of 3 or greater

Exclusion Criteria:

* Hematological abnormalities
* Heart rate < 50 or > 90 bpm when resting for 5 minutes
* Family history of long QT syndrome
* History of tachyarrhythmia
* History of conduction abnormality i.e., PR > 200 msec, 2nd or 3rd degree AV block, complete left or right branch bundle block, pre-excitation syndrome
* Uncontrolled or unstable angina pectoris; history of myocardial infarction within the previous 12 months
* Known history of congestive heart failure
* History of percutaneous coronary intervention (PCI) or cardiac ablation
* History of stroke or transient ischemic attack (TIA)
* Implanted cardiac pacemaker or defibrillator
* History of malignancy of any organ system
* Current guttate, generalized erythrodermic, or pustular psoriasis
* Current drug associated psoriasis

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plaque psoriasis as assessed by PASI response or PASI 75 (a patient that has an improvement from baseline PASI of at least 75%) | to 12 weeks treatment

SECONDARY OUTCOMES:
ECG and laboratory parameters, rates of AEs, and percentage of patients requiring interruption or discontinuation of study drug due to AEs | up to 12 weeks treatment
change in PASI and Investigator's Global Assessment (IGA) of psoriasis in patients receiving AEB071 compared with placebo | up to 12 weeks treatment
disease recurrence (PASI, IGA) and the effect of treatment withdrawal (including AEs) in the treatment-free Follow-up Period | in the treatment-free Follow-up Period

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- United States (10):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - Belleair Research Center, LLC, Pinellas Park, Florida
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Dermatology Specialists, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Central Dermatology, St Louis, Missouri
  - Palmetto Clinical Trial Services, Greenville, South Carolina
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce & Associates, PA, Houston, Texas
  - Virginia Clinical Research, Norfolk, Virginia
- Argentina (2):
  - Novartis Investigative site, Buenos Aires
  - Novartis Investigative site, Mendoza
- Australia (4):
  - Novartis Investigative site, Benowa
  - Novartis Investigative site, Carlton
  - Novartis Investigative site, Kogarah
  - Novartis Investigative site, Parkville
- Belgium (3):
  - Novartis Investigative site, Brussels
  - Novartis Investigative site, Edegem
  - Novartis Investigative site, Liège
- Germany (8):
  - Novartis Investigative site, Berlin
  - Novartis Investigative site, Bonn
  - Novartis Investigative site, Erlangen
  - Novartis Investigative site, Frankfurt
  - Novartis Investigative site, Hamburg
  - Novartis Investigative site, Kiel
  - Novartis Investigative site, Leipzig
  - Novartis Investigative site, Regensburg
- Novartis Investigative Site, Guatemala City, Guatemala
- Italy (5):
  - Novartis Investigative site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Siena
  - Novartis Investigative Site, Verona
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Manisa
- United Kingdom (3):
  - Novartis Investigative site, Nuneaton
  - Novartis Investigative site, Salford
  - Novartis Investigative site, Southampton

REFERENCES:
- See also: Results for CAEB071C2201 from the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6743